CLINICAL TRIAL: NCT00482664
Title: A Phase 2a Multi-Centre, Double Blind, Placebo Controlled Cross-Over Trial To Investigate The Efficacy, Safety And Toleration Of CP-866,087 In Pre-Menopausal Women Diagnosed With Female Sexual Arousal Disorder (FSAD).
Brief Title: The Efficacy, Safety And Toleration Of CP-866,087 In Pre-Menopausal Women With Female Sexual Arousal Disorder.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A5051017
Record Dates: First submitted 2007-06-01; First posted 2007-06-05 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Sexual Dysfunction, Physiological
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — CP-866,087

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- 1 mg (Experimental)
  Interventions: Drug: CP-866,087
- 10 mg (Experimental)
  Interventions: Drug: CP-866,087
- 3 mg (Experimental)
  Interventions: Drug: CP-866,087
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CP-866,087 — Tablets for oral administration
  Arms: 1 mg
Drug: CP-866,087 — Tablets for oral administration
  Arms: 10 mg
Drug: CP-866,087 — Tablets for oral administration
  Arms: 3 mg
Drug: Placebo — Tablets for oral administration
  Arms: Placebo

SUMMARY:
CP-866,087 is a non-hormonal compound, acting on the central nervous system, which has been shown in animal models to restore sexual function.

ELIGIBILITY:
Inclusion Criteria:

* healthy pre-menopausal women
* primary female sexual arousal disorder causing distress
* on stable use of oral contraceptives

Exclusion Criteria:

* any other significant disease causing Female Sexual Dysfunction including psychiatric disease
* subjects on drugs known to cause Female Sexual Dysfunction
* subjects who have given birth in the last 12 months or who are planning to become pregnant during the study

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Diary events, including Satisfactory Sexual Experiences (SSEs) over 6 weeks. | 6 weeks
Score in Abbreviated Sexual Function Questionnaire after 6 weeks of treatment. | 6 weeks

SECONDARY OUTCOMES:
Exit interview at end of study. Meaningful Benefit Question at end of study. | End of study
Measure of Female Sexual Distress questionnaire after 6 weeks of treatment. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (11):
- Australia (2):
  - Pfizer Investigational Site, Dulwich, South Australia
  - Pfizer Investigational Site, Nedlands, Western Australia
- Denmark (3):
  - Pfizer Investigational Site, Aarhus C
  - Pfizer Investigational Site, Kobenhavn OE
  - Pfizer Investigational Site, Odense C
- Pfizer Investigational Site, Oslo, Norway
- South Africa (2):
  - Pfizer Investigational Site, Westville, KwaZulu-Natal
  - Pfizer Investigational Site, Pretoria
- Sweden (3):
  - Pfizer Investigational Site, Lund
  - Pfizer Investigational Site, Skövde
  - Pfizer Investigational Site, Stockholm

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5051017&StudyName=The%20Efficacy%2C%20Safety%20And%20Toleration%20Of%20CP-866%2C087%20In%20Pre-Menopausal%20Women%20With%20Female%20Sexual%20Arousal%20Disorder.